CLINICAL TRIAL: NCT00797056
Title: Pilot Study of Stem Cell Mobilization by G-CSF to Treat Severe Peripheral Artery Disease (STEMPAD Trial)
Brief Title: Stem Cell Mobilization by G-CSF to Treat Severe Peripheral Artery Disease
Acronym: STEMPAD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-0043 / 201106083
Record Dates: First submitted 2008-11-20; First posted 2008-11-25 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Peripheral Vascular Diseases
Keywords: G-CSF; angiogenesis; endothelial progenitor cell; limb ischemia; revascularization
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF (Experimental)
  Interventions: Drug: G-CSF; Drug: Aspirin; Drug: Clopidogrel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: G-CSF — G-CSF 5 mcg/kg/day SQ daily for 10 days
  Other Names: Filgrastim; Neupogen
  Arms: G-CSF
Drug: Placebo — Saline SQ daily for 10 days
  Other Names: NaCl
  Arms: Placebo
Drug: Aspirin — Aspirin 75 mg/day for 14 days
  Other Names: acetylsalicylate
Drug: Clopidogrel — Clopidogrel 75mg/day daily for 14 days
  Other Names: Plavix

SUMMARY:
This study is designed to test the use of G-CSF in peripheral vascular disease. The investigators hypothesize that mobilization of angiogenic cells into the blood by granulocyte colony stimulating factor (G-CSF) may stimulate the formation of new blood vessels and result in a sustained improvement in blood flow in patients with severe peripheral arterial disease.

DETAILED DESCRIPTION:
One fourth of patients with peripheral artery disease (PAD) of the lower extremities have severe symptomatic disease and 1-2% have critical limb ischemia (CLI). In patients with CLI, the risk of limb amputation at 1 year is 50%. In addition, patients with CLI often have rest pain, non-healing ulcers and severe limitations of ambulation. Revascularization procedures, including bypass surgery, percutaneous transluminal angioplasty and angioplasty with stenting, are currently the only treatment options. However, many patients are not eligible for a revascularization procedure due to small vessel disease or coexisting medical problems. Moreover, restenosis rates are high.

There is currently no effective non-invasive treatment for critical limb ischemia. We hypothesize that mobilization of angiogenic cells into the blood by granulocyte colony stimulating factor (G-CSF) may stimulate angiogenesis in areas of ischemia and result in a sustained improvement in blood flow in patients with severe PAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have critical limb ischemia secondary to PAD, as defined by the presence of a non-healing ulcer, rest pain, or dry gangrene.
* Patients must have a toe pressure ≤ 30 mm Hg.
* Patients must be ≥18 years old.
* Patient must be able to self-administer a daily subcutaneous injection or have a caregiver who is able to administer a daily subcutaneous injection.
* Patients must be taking or have no absolute contraindication to taking aspirin and clopidogrel. If they are not currently taking aspirin, they must be willing to take aspirin (81 mg daily) and clopidogrel (75 mg daily) for 14 days starting on the first day of G-CSF treatment.
* After being informed of the treatment involved, patients must give written consent. The patient should not have any serious medical or psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment. A built-in period of one week from discussion of the trial and initiation of the trial will be mandatory for enrollment.

Exclusion Criteria:

* Patients with transmetatarsal or higher amputations in the affected limb are excluded.
* Patients who are candidates for a revascularization procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Major limb amputation rate as defined by amputations of the limb that are transmetarsal and higher | 1 year

SECONDARY OUTCOMES:
Toe pressure index | Up to 1 year
  Toe brachial index (TBI) and is a calculation based on the systolic blood pressures of the arm and the systolic blood pressures of the toes. The examination is performed with a photoplethysmograph (PPG) infrared light sensor and a very small blood pressure cuff placed around the toe.
  The arm and big toe systolic blood pressure measurements are recorded. Then the big toe systolic pressures are divided by the highest arm pressure to establish an TBI measurement for each leg. A TBI of .75 or greater is consider normal.
Ankle-brachial index | Up to 1 year
  * The Ankle Brachial Index (ABI or ABPI) is the ratio of the blood pressure in the lower legs to the blood pressure in the arms. Compared to the arm, lower blood pressure in the leg is an indication of blocked arteries (peripheral vascular disease or PVD). The ABI is calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressures in the arm.
  * A normal resting ankle-brachial index is 1 or 1.1.
  A resting ankle-brachial index of less than 1 is abnormal. If the ABI is:
  * Less than 0.95, significant narrowing of one or more blood vessels in the legs is indicated.
  * Less than 0.8, pain in the foot, leg, or buttock may occur during exercise (intermittent claudication).
  * Less than 0.4, symptoms may occur when at rest.
  * 0.25 or below, severe limb-threatening peripheral artery disease is probably present.
Ulcer healing as measured by surface area and depth | Up to 1 year
  * Skin ulcerations should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeat measurements. A maximum of 3 ulcers on each lower extremity will be followed.
  * An average of the longest diameter for all ulcerations will be calculated and reported as the baseline average longest diameter. The baseline average will be used as reference by which to characterize the ulcerations.
Improvement in rest pain as measured by the Vascular Quality of Life Questionnaire | Up to 1 year
  -25 questions including questions in activity, symptom, pain, emotional, and social domains.
  Each question has seven choices ranging from "All" to "None"
  * Each domain is scored 1-7=the total of domain item scores divided by the number of questions in the domain.
  * The total score is is also scored 1-7=the total of all the item scores divided by 25.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Geraghty, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu